CLINICAL TRIAL: NCT04782778
Title: Comparison of Ultrasound-Guided Supraclavicular and Costoclavicular Brachial Plexus Blocks in Pediatric Patients Undergoing Unilateral Upper Exremity Surgery: A Randomized Controlled Double-Blinded Study
Brief Title: Comparison of Supraclavicular and Costoclavicular Brachial Plexus Blocks in Pediatrics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Meltem Savran Karadeniz, Associate Professor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: 2020/46
Record Dates: First submitted 2021-03-02; First posted 2021-03-04 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Anesthesia, Local; Postoperative Pain
Keywords: Postoperative Analgesia; Upper Extremity Surgery; Supraclavicular Block; Costoclavicular Block; Brachial Plexus Block; Ultrasound Guidance
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: RANDOMISED DOUBLE BLINDED INTERVENTIONAL
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Costoclavicular Block (Active Comparator): US-guided lateral approach costoclavicular block with 1 mg/kg Bupivacaine (%0,25)
  Interventions: Drug: Bupivacaine 0.25% Injectable Solution
- Ultrasound Guided Supraclavicular Block (Active Comparator): US-guided supraclavicular block with 1 mg/kg Bupivacaine (%0,25)
  Interventions: Drug: Bupivacaine 0.25% Injectable Solution

INTERVENTIONS:
Drug: Bupivacaine 0.25% Injectable Solution — 1 mg/kg Bupivacaine (0.25%)
  Other Names: Marcaine

SUMMARY:
In upper extremity surgeries, the brachial plexus block can be performed with different techniques at various levels depending on the proximal and distal level of the surgery.

As an alternative to the infraclavicular brachial plexus block, which has been used for many years and which we routinely perform to every pediatric patient under general anesthesia; Costoclavicular block is recommended due to its advantages such as short application time, single injection and sufficient ultrasound imaging, and its use is becoming widespread. There are studies comparing these two methods. However in this study, we aim to compare the postoperative analgesic effects of US-guided costoclavicular technique with US-guided supraclavicular technique, which is more common for many years and is performed 2-3 cm proximal to the costoclavicular block area.

During the block application, the US imaging time, the difficulty level of needle imaging, the number of maneuvers required to reach the target image, whether additional maneuvers are required according to the local anesthetic distribution, the success of the block and the duration of the surgery, the total application time of the block and the duration of general anesthesia will be recorded. Mean arterial pressure and heart rate will be recorded at 30-minute intervals during the surgery. Standardized for pediatric patients The FLACC and Wong-Baker pain scores will be followed first 24 hours after surgery. The patient will be examined for pain, motor and sensation, and analgesic doses will be recorded if used. Time to first pain identification, duration of sleep, patient and surgeon satisfaction will be recorded.

The rarely onset of hemidiaphragmatic paralysis during supraclavicular block reduces its use. Costoclavicular block could be a safe and effective alternative. One of our seconder objectives is to assess the incidence of hemidiaphragmatic paralysis following ultrasound-guided supraclavicular block and compare it to that of costoclavicular block. For this purpose diaphragmatic excursion is visualized by M-mode ultrasonography 30 minutes after extubation. In B-mode, the diaphragm thickness measurement at the end of expiratory and inspiratory end is recorded and the diaphragm thickness fraction is calculated. Absence of diaphragmatic excursion during a sniff test or sighing defined the hemidiaphragmatic paralysis.

DETAILED DESCRIPTION:
Peripheral nerve blocks; It is widely used in daily practice for anesthesia or as a part of multimodal analgesia in most surgical procedures. In upper extremity surgeries, the brachial plexus block can be performed with different techniques at various levels depending on the proximal and distal level of the surgery. In this study, the aim is to compare postoperative analgesic effects of these two ultrasound-guided techniques in pediatric patients.

As an alternative to the infraclavicular brachial plexus block, which has been used for many years and which we routinely perform to every pediatric patient under general anesthesia; Costoclavicular block is recommended due to its advantages such as short application time, single injection and sufficient ultrasound imaging, and its use is becoming widespread. There are studies comparing these two methods. However, we aim to compare the costoclavicular technique with the supraclavicular technique, which is more common for many years and is performed 2-3 cm proximal to the costoclavicular block area. Thus demonstrate the safety of upper extremity blocks, which is an important part of multimodal analgesia, and to determine the most ideal technique in the pediatric patient group who will undergo upper extremity surgery.

During the block application, the US imaging time, the difficulty level of needle imaging, the number of maneuvers required to reach the target image, whether additional maneuvers are required according to the local anesthetic distribution, the success of the block and the duration of the surgery, the total application time of the block and the duration of general anesthesia will be recorded. Mean arterial pressure and heart rate will be recorded at 30-minute intervals during the surgery. Standardized for pediatric patients The FLACC and Wong-Baker pain scores will be followed first 24 hours after surgery. The patient will be examined for pain, motor and sensation, and analgesic doses will be recorded if used. Time to first pain identification, duration of sleep, patient and surgeon satisfaction will be recorded.

The rarely onset of hemidiaphragmatic paralysis during supraclavicular block reduces its use. Costoclavicular block could be a safe and effective alternative. One of our seconder objectives is to assess the incidence of hemidiaphragmatic paralysis following ultrasound-guided supraclavicular block and compare it to that of costoclavicular block. For this purpose diaphragmatic excursion is visualized by M-mode ultrasonography 30 minutes after extubation. In B-mode, the diaphragm thickness measurement at the end of expiratory and inspiratory end is recorded and the diaphragm thickness fraction is calculated. Absence of diaphragmatic excursion during a sniff test or sighing defined the hemidiaphragmatic paralysis.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing unilateral upper extremity surgery (distal midhumerus).
* ASA(American Society of Anesthesiology) 1-3
* Receiving family consent from the parents that they accept regional analgesia

Exclusion Criteria:

* Parents refusal
* Infection on the local anesthetic application area
* Infection in the central nervous system
* Coagulopathy
* Brain tumors
* Known allergy against local anesthetics
* Anatomical difficulties
* Syndromic patient

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Total block application time | Up to 15 minutes
  Total block application time from the needle's entrance to the exit from the skin

SECONDARY OUTCOMES:
Ideal USG guided brachial plexus cords visualization/needle pathway planning time | Up to 15 minutes
  Practitioner's ideal image acquisition time
Needle tip and shaft imaging visualization | Up to 15 minutes
  Likert scale: 1-5 (1:very hard 5:very easy)
Number of needle maneuvers | Up to 15 minutes
  Number of needle maneuvers according to local anesthetic distribution
Total procedure difficulty according to the anesthesiologist | Up to 15 minutes
  Likert Scale: 1-5 (1:very hard 5:very easy)
Patient number requiring rescue analgesics | Intraoperative 2-4 hours
  If a ≥ 20% increase above preinduction values in MAP or HR was observed during the perioperative period, additional fentanyl dose (1 μg/kg) was applied intravenously.
Face, Legs Activity, Cry, Consolability (FLACC) scores | Up to 24 hours
  It corporates five categories of behavior, each scored on 0-2 point scale so that total score ranges from 0 to 10. Total scores of 0-3 is defined as mild or no pain, 4-7 as moderate, and 8-10 as severe pain.
Wong Baker FACES scale | Up to 24 hours
  The scale shows a series of faces ranging from a happy face at 0, or "no hurt", to a crying face at 10, which represents "hurts like the worst pain imaginable"
Motor blockade physical examination | Up to 24 hours
  Each nerve scored on 0-2 point scale so that total score ranges from 0 to 8. Total scores of 0 point is defined as absent motor blockade (full movement); 1 point as partial blockade (able to free movement only) or 2 point as complete blockade (unable to move). (Separately for these four nerves; N. Medianus, N. ulnaris, N. radialis and N. musculocutaneous).
Sensorial blockade physical examination | Up to 24 hours
  Each nerve scored on 0-2 point scale with pinprick test so that total score ranges from 0 to 8. Total scores of 0 point is defined as absent sensorial blockade (feels pain), 1 point as partial blockade (feels touch) or 2 point as complete blockade (no sense). (Separately for these four nerves; N. Medianus, N. ulnaris, N. radialis and N. musculocutaneous).
Complications/side effects | Up to first week
  Vascular puncture, hematoma, pleura puncture, infections, phrenic nerve paralysis
Incidence of symptomatic/asymptomatic postprocedural phrenic nerve paralysis | Up to 2 hours
  Diaphragmatic excursion is visualized by M-mode ultrasonography 30 minutes after extubation. In B-mode, the diaphragm thickness measurement at the end of expiratory and end of inspiratory is recorded and the diaphragm thickness fraction is calculated.
Time to postoperative first pain | Up to 24 hours
  Time to first analgesic
Patient number who require additional analgesic | Up to 24 hours
  Number of patients who require IV morphine (0.03 mg/kg) and paracetamol
Duration of sleep | Up to 24 hours
  Total hours of sleep first day
Family satisfaction | Up to 24 hours
  Satisfaction score: 0: very unsatisfied, 3: very satisfied
Surgeon satisfaction | Up to 24 hours
  Satisfaction score: 0: very unsatisfied, 3: very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Meltem Savran Karadeniz, Assoc.Prof., Principal Investigator — Istanbul University
Locations (1):
- Istanbul University, Istanbul, Fatih, Turkey (Türkiye)

REFERENCES:
- [Background] Songthamwat B, Karmakar MK, Li JW, Samy W, Mok LYH. Ultrasound-Guided Infraclavicular Brachial Plexus Block: Prospective Randomized Comparison of the Lateral Sagittal and Costoclavicular Approach. Reg Anesth Pain Med. 2018 Nov;43(8):825-831. doi: 10.1097/AAP.0000000000000822. PMID 29923950
- [Background] Grape S, Pawa A, Weber E, Albrecht E. Retroclavicular vs supraclavicular brachial plexus block for distal upper limb surgery: a randomised, controlled, single-blinded trial. Br J Anaesth. 2019 Apr;122(4):518-524. doi: 10.1016/j.bja.2018.12.022. Epub 2019 Jan 31. PMID 30857608
- [Background] Sivashanmugam T, Maurya I, Kumar N, Karmakar MK. Ipsilateral hemidiaphragmatic paresis after a supraclavicular and costoclavicular brachial plexus block: A randomised observer blinded study. Eur J Anaesthesiol. 2019 Oct;36(10):787-795. doi: 10.1097/EJA.0000000000001069. PMID 31397702
- [Background] Luo Q, Yao W, Chai Y, Chang L, Yao H, Liang J, Hao N, Guo S, Shu H. Comparison of ultrasound-guided supraclavicular and costoclavicular brachial plexus block using a modified double-injection technique: a randomized non-inferiority trial. Biosci Rep. 2020 Jun 26;40(6):BSR20200084. doi: 10.1042/BSR20200084. PMID 32441302